CLINICAL TRIAL: NCT04242381
Title: Short Term Effect Of Kinesiotaping on Pain, Functionality, and Ultrasound Parameters In Patients With Shoulder Impingement Syndrome: A Randomized Sham-Controlled Study
Brief Title: Short Term Effect of Kinesiotaping In Patients With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kars State Hospital (Other)
Responsible Party: Principal Investigator, Fatih Bagcier, Principal Investigator, Kars State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HNEAH-KAEK 2016/269
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Kinesiotape; Exercise; Ultrasound
Keywords: Kinesiotape; exercise; ultrasound
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A Randomized Sham-Controlled Study
Who Masked: Investigator
Masking Description: All participants were assessed by the same clinician (F.B) at the baseline and at the two week after completing the interventions by visual analog scale (VAS), range of motion (ROM) and Disabilities of the Arm, Shoulder and Hand Questionnaire (Q-DASH). KT and sham-KT applications were made by same clinician (N.M). For ultrasnogohraphic (US) measurements, the participants were sent to a clinician (D.G.K) who was blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Cold application, Kinesiotaping treatment (Experimental): Cold application: At the beginning of each treatment session, gel ice packs were wrapped in a damp towel and applied to the patients' shoulder joints for 20 minutes.
  Kinesiotaping application: KT was applied to the deltoid muscle using the inhibition and mechanical correction technique and to the supraspinatus muscle using the inhibition technique (2 sessions with a 5-day interval).
  Interventions: Other: Cold Application; Other: Kinesiotaping Application
- Group 2: Cold application, EX treatment (Experimental): EX treatment was administered for 10 days with 3 sessions/day. A triphasic exercise program was administered to the patients. Exercise was administered twice a week under supervision; however, the patients were advised to exercise at home on the other days with 20 repetitions of each exercise. The patients were followed up via telephone to make sure they were adhering to their exercise programs.
  Interventions: Other: Cold Application; Other: Exercise treatment
- Group 3: Cold application, sham-KT treatment (Sham Comparator): Sham-KT was applied in 10 cm I-shaped stripes on the sagittal plane over the acromioclavicular joint without stretching and on the transverse plane distal to the deltoid area. The kinesiotape was applied twice for five days with 2-day intervals
  Interventions: Other: Cold Application; Other: Sham Kinesio taping application

INTERVENTIONS:
Other: Cold Application — At the beginning of each treatment session, gel ice packs were wrapped in a damp towel and applied to the patients' shoulder joints for 20 minutes.
Other: Kinesiotaping Application — KT was applied to the deltoid muscle using the inhibition and mechanical correction technique and to the supraspinatus muscle using the inhibition technique (2 sessions with a 5-day interval)
  Arms: Group 1: Cold application, Kinesiotaping treatment
Other: Exercise treatment — EX treatment was administered for 10 days with 3 sessions/day. A triphasic exercise program was administered to the patients. Before starting the exercise program, the patients were instructed to not perform the movements exceeding 90° overhead. The exercise program was initiated using codman pendulum, passive joint motion range (with a 1-m stick), and posterior capsule stretching exercise. Shoulder wheel, finger ladder, and shoulder strengthening exercise with theraband were added to the exercise programs of patients with full or near total range of motion and pain relief. Exercise was administered twice a week under supervision; however, the patients were advised to exercise at home on the other days with 20 repetitions of each exercise. The patients were followed up via telephone to make sure they were adhering to their exercise programs.
  Arms: Group 2: Cold application, EX treatment
Other: Sham Kinesio taping application — Sham-KT was applied in 10 cm I-shaped stripes on the sagittal plane over the acromioclavicular joint without stretching and on the transverse plane distal to the deltoid area. The kinesiotape was applied twice for five days with 2-day intervals
  Arms: Group 3: Cold application, sham-KT treatment

SUMMARY:
We aimed to investigate the effect of kinesiotaping on pain, functionality and ultrasound parameters in patients with shoulder impingement syndrome (SIS).

DETAILED DESCRIPTION:
A total of 75 patients with SIS were randomly classified into the following three groups: kinesiotaping (KT), exercise (EX) and sham-kinesiotaping (sham-KT). Each group was underwent two weeks treatment program. The patients were then evaluated in terms of pain analyzed using the visual analog scale (VAS), joint range of motion, Quick-Disabilities of the Arm, Shoulder and Hand (Q-DASH) questionnaire before and after treatment. In addition, supraspinatus tendon (SsT) thickness and acromiohumeral distance (AHD) parameters were measured using ultrasonography (US). All parameters were measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* at least three positive results in the Hawkins-Kennedy, Neer, empty can, drop-arm, and lift-off tests
* magnetic resonance imaging findings
* age between 45 and 70 years

Exclusion Criteria:

* Patients who received physical therapy for the shoulder region within the past three months or those with a history of injections to the shoulder joint,
* cervical pathologies,
* clinical conditions accompanied by neuromotor or sensory dysfunction,
* history of malignancy,
* pregnancies,
* partial or total rupture in the supraspinatus tendon,
* adhesive capsulitis,
* diabetes or chronic liver, or kidney failure

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Level | 4 weeks
  The severity of shoulder pain (resting, activity, and night pain) in the patients was evaluated through the VAS score. A VAS score of 0 represented no pain, whereas a score of 10 represented the most severe pain; the patients were asked to mark the average severity of the pain they felt during the past week and the marked point was measured using a centimeter ruler and recorded.
Functional Status | 4 weeks
  Quick-Disabilities of the Arm, Shoulder and Hand (Q-DASH) questionnaire: This questionnaire comprises three sections. The first section comprises 30 items: 21 items assess the patient's difficulties in performing daily activities, 5 assess symptoms (pain, activity-related pain, tingling, stiffness, and weakness), and each of the remaining 4 items assesses social function, work, sleep, and self-confidence. All items are rated on a 5-point Likert-type scale (1, no difficulty; 2, mild difficulty; 3, moderate difficulty; 4, extreme difficulty; 5, cannot perform at all). The total score possible through this questionnaire ranges from 0 to 100 (0, no disability; 100, maximum disability). Furthermore, Turkish reliability and validity have been performed for this questionnaire.
Joint range of motion measurements | 4 weeks
  Flexion (FLX), abduction (ABD), internal rotation (IR) and external rotation (ER) were measured using a goniometer (saehan gonıometer - plastıc).
Ultrasonography | 4 weeks
  US was performed using a 7.5-mHz linear probe in the B mode (Mindray-China). Supraspinatus tendon (SsT) thickness was measured at three different points (10, 15, and 20 mm) lateral to the tendon after identifying the biceps tendon in the transverse section and the average of measurements was recorded. Acromiohumeral distance (AHD) was assessed by linearly measuring the distance between the inferior of the acromion from the anterior of the shoulder and the superior of the humeral head

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No